CLINICAL TRIAL: NCT03173326
Title: Randomized Controlled Trial Evaluating Patient Satisfaction and Postoperative Analgesia Between Subarachnoid Block With 2-chloroprocaine Versus General Anesthesia for Knee Arthroscopy
Brief Title: Patient Satisfaction and Postoperative Analgesia Between Subarachnoid Block With 2-chloroprocaine Versus General Anesthesia for Knee Arthroscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing changes at site. No longer feasible at site.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jenna Walters, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170741
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Knee Arthroscopy; General Anesthesia; Subarachnoid Block
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subarachnoid block (Experimental)
  Interventions: Procedure: Subarachnoid block
- General anesthesia (Active Comparator)
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: General anesthesia — General anesthesia will be delivered per standard procedure. General anesthesia will include induction with propofol 1-3mg/kg followed by placement of a laryngeal mask airway with maintenance anesthesia of sevoflurane 0.5-1 minimum alveolar concentration (MAC).
  Arms: General anesthesia
Procedure: Subarachnoid block — Neuraxial anesthesia will be performed at the L2-3 or L3-4 interspace with a 25-gauge Whitacre needle in the sitting position. After free flow of cerebrospinal fluid (CSF), 40-45mg of 2-chloroprocaine will be injected based on patient's height and discretion of attending anesthesiologist, needle withdrawn and the patient placed supine.
  Arms: Subarachnoid block

SUMMARY:
The study evaluates the efficacy of two different anesthetic techniques in patients undergoing unilateral knee arthroscopy. Participants will be randomized to receive either subarachnoid block with 2-chloroprocaine or general anesthesia plus intravenous fentanyl.

DETAILED DESCRIPTION:
The study evaluates the efficacy of two different anesthetic techniques in patients undergoing unilateral knee arthroscopy. Participants will be randomized to receive either subarachnoid block with 2-chloroprocaine or general anesthesia plus intravenous fentanyl. The study evaluates pain scores, opioid utilization and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA physical status classification of I, II, or III
* Patients without a current diagnosis of chronic pain or chronic opioid use for > 1-month prior to knee arthroscopy
* Patients who are scheduled to undergo unilateral knee arthroscopy
* Patients do not have a contraindication to receiving regional anesthesia

Exclusion Criteria:

* Preexisting sensory or motor deficit in operative extremity
* Patients with a contraindication to general anesthesia
* Patient undergoing meniscal or ligamentous repair

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Pain score | Discharge from post anesthesia care unit (PACU) (usually one hour)
  Pain score measured with a patient reported 11 point Numeric Rating Pain Scale with 0 indicating no pain and 10 indicating worst pain imaginable.
Pain score | Post operative day one
  Pain score measured with a patient reported 11 point Numeric Rating Pain Scale with 0 indicating no pain and 10 indicating worst pain imaginable.
Pain score | One month postoperatively
  Pain score measured with a patient reported 11 point Numeric Rating Pain Scale with 0 indicating no pain and 10 indicating worst pain imaginable.
Pain score | Three months postoperatively
  Pain score measured with a patient reported 11 point Numeric Rating Pain Scale with 0 indicating no pain and 10 indicating worst pain imaginable.
Opioid utilization | Surgical completion to PACU discharge (usually one hour)
  Opioid utilization based on amount of opioid medications administered
Opioid utilization | Postoperative day one
  Opioid utilization based on number of pain pills taken
Opioid utilization | One month postoperatively
  Opioid utilization based on average number of pain pills taken per day
Opioid utilization | Three months postoperatively
  Opioid utilization based on average number of pain pills taken per day

SECONDARY OUTCOMES:
Patient satisfaction with anesthetic | 24 hours after PACU discharge
  Patient satisfaction with anesthetic based on 10-item patient satisfaction survey validated for regional and general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Walters, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No